CLINICAL TRIAL: NCT01537887
Title: A Placebo- and Positive-Controlled Study of the Effect of LY2484595 on QT Interval in Healthy Subjects
Brief Title: A Study of LY2484595 on the Electrical Activity of the Heart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 11947; I1V-MC-EIAK (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — evacetrapib; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Administered orally once daily for 10 days during 1 of the 3 crossover periods, separated by at least a 14-day washout period.
  Interventions: Drug: Placebo
- 1200 milligrams (mg) LY2484595 (Experimental): Administered orally once daily for 10 days during 1 of the 3 crossover periods, separated by at least a 14-day washout period.
  Interventions: Drug: LY2484595
- 400 mg Moxifloxacin (Active Comparator): Positive control, unblinded treatment administered orally once during 1 of 3 crossover periods, separated by at least a 14-day washout period.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: LY2484595 — Administered orally once daily for 10 days.
  Arms: 1200 milligrams (mg) LY2484595
Drug: Placebo — Administered orally once daily for 10 days.
  Arms: Placebo
Drug: Moxifloxacin — Single dose administered orally.
  Arms: 400 mg Moxifloxacin

SUMMARY:
The purpose of this study is to evaluate the effect on the electrical activity of the heart as measured by an electrocardiogram (ECG) after dosing with 10 days of LY2484595 compared to 10 days of placebo in relation to a single dose of moxifloxacin. Information about any side effects that occur will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Body mass index (BMI) of 18.5 to 29 kilograms per square meter (kg/m²)
* Reliable and willing to be available for the duration of the study and are willing to follow study procedures
* Provided written informed consent

Exclusion Criteria:

* Known allergies to LY2484595 or moxifloxacin
* Personal or family history of long QT syndrome, heart failure, or low blood potassium (hypokalemia) a family history of sudden death, or unexplained syncope within the last year
* Positive findings on urinary drug screening
* Cigarette smokers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to 1 of 6 treatment sequences in a crossover design with 3 treatments; 1200 mg LY2484595, then placebo, then moxifloxacin. There was a washout period of ≥14 days between each dose. Participants were dosed 3 times during the entire study.
Groups:
- Sequence 1: Placebo or 1200 milligrams (mg) LY2484595 administered orally twice daily for 10 days, or 400 mg moxifloxacin single oral dose on Day 1 during 1 of the 3 crossover periods. There was at least 14 days washout between consecutive dosing periods.
  Sequence 1 (ABC): LY248495, then placebo, then moxifloxacin
- Sequence 2: Placebo or 1200 mg LY2484595 administered orally twice daily for 10 days, or 400 mg moxifloxacin single oral dose on Day 1 during 1 of the 3 crossover periods. There was at least 14 days washout between consecutive dosing periods.
  Sequence 2 (BCA): placebo, then moxifloxacin, then LY2484595
- Sequence 3: Placebo or 1200 mg LY2484595 administered orally twice daily for 10 days, or 400 mg moxifloxacin single oral dose on Day 1 during 1 of the 3 crossover periods. There was at least 14 days washout between consecutive dosing periods.
  Sequence 3 (CAB): moxifloxacin, then LY2484595, placebo
- Sequence 4: Placebo or 1200 mg LY2484595 administered orally twice daily for 10 days, or 400 mg moxifloxacin single oral dose on Day 1 during 1 of the 3 crossover periods. There was at least 14 days washout between consecutive dosing periods.
  Sequence 4 (CBA): moxifloxacin, then placebo, then LY2484595
- Sequence 5: Placebo or 1200 mg LY2484595 administered orally twice daily for 10 days, or 400 mg moxifloxacin single oral dose on Day 1 during 1 of the 3 crossover periods. There was at least 14 days washout between consecutive dosing periods.
  Sequence 5 (ACB): LY2484595, then moxifloxacin, then placebo
- Sequence 6: Placebo or 1200 mg LY2484595 administered orally twice daily for 10 days, or 400 mg moxifloxacin single oral dose on Day 1 during 1 of the 3 crossover periods. There was at least 14 days washout between consecutive dosing periods.
  Sequence 6 (BAC): placebo, then LY2484595, then moxifloxacin
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 12 | 12 | 12 | 12 | 12 | 12
Received at Least 1 Dose of Study Drug | 12 | 12 | 11 | 12 | 12 | 12
Completed | 12 | 12 | 11 | 12 | 11 | 11
Not Completed | 0 | 0 | 1 | 0 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Did not receive treatment | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 12 | 12 | 11 | 12 | 11 | 11
Completed | 12 | 11 | 11 | 12 | 11 | 11
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 12 | 11 | 11 | 12 | 11 | 11
Completed | 12 | 10 | 10 | 12 | 11 | 11
Not Completed | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants received at least one dose of study drug.
Groups:
- All Participants: Placebo or 1200 mg LY2484595 administered orally once daily for 10 days, or 400 mg moxifloxacin single oral dose on Day 1 during 1 of the 3 crossover periods. There was at least 14 days washout between consecutive dosing periods.
Arm/Group | All Participants
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 52
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 17
  White | 53
  More than one race | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 71

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 10 in QT Interval Corrected for Heart Rate (QTc) for LY2484595 Versus Placebo
Description: Data were collected using a 12-lead electrocardiogram (ECG). The QT interval is the time between the start of the Q wave and the end of the T wave in the cardiac electrical cycle and corrected for heart rate. Population-corrected QT interval (QTcP) formula: QTcP = QT / RR^ß, where ß is the population correction factor.
Time Frame: Predose of Day 1, Day 10
Population: All participants who received at least one dose of study drug and had both baseline and post-baseline ECG measurements on Day 10.
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Groups:
- Placebo: Administered orally once daily for 10 days during 1 of the 3 crossover periods. There was at least 14 days washout between consecutive dosing periods.
- LY2484595: 1200 milligrams (mg) LY2484595 administered orally once daily for 10 days during 1 of the 3 crossover periods. There was at least 14 days washout between consecutive dosing periods.
Arm/Group | Placebo | LY2484595
Number analyzed (Participants) | 68 | 69
milliseconds (msec)
  4-hour postdose on Day 10: number analyzed (Participants) | 68 | 68
  4-hour postdose on Day 10 | -2.7 (7.5) | -4.6 (8.5)
  6-hour postdose on Day 10: number analyzed (Participants) | 67 | 69
  6-hour postdose on Day 10 | -2.0 (7.7) | -1.1 (8.5)

2. Secondary Outcome: Pharmacokinetics: Maximum Drug Concentration (Cmax) of LY2484595 During One Dosing Interval at Steady State
Time Frame: Predose, 1, 2, 3, 4, 6, 12, 24, 72, and 168 Hours Postdose
Population: Participants who received at least one dose of LY2484595 and had pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | LY2484595
Number analyzed (Participants) | 69
nanograms/milliliter (ng/mL) | 5270 (65)

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY2484595 During One Dosing Interval at Steady State
Time Frame: Predose, 1, 2, 3, 4, 6, 12, 24, 72, and 168 Hours Postdose
Population: Participants who received at least one dose of LY2484595 and had pharmacokinetic data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Arm/Group | LY2484595
Number analyzed (Participants) | 69
nanograms*hour/milliliter (ng*h/mL) | 48300 (49)

4. Secondary Outcome: Percentage Change From Baseline to Day 11 in Fasting Lipids and Apolipoproteins
Time Frame: Baseline, Day 11
Population: All participants who received at least one dose of study drug and had both baseline and post-baseline lipid or apolipoprotein (Apo) measurements on Day 11.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Placebo | LY2484595
Number analyzed (Participants) | 68 | 69
percentage change
  High-density lipoprotein cholesterol (HDL-C) | -8 (15) | 112 (37)
  Low-density lipoprotein cholesterol (LDL-C) | 9 (17) | -35 (16)
  Apo-A1 | -9 (13) | 32 (18)
  Apo-B: number analyzed (Participants) | 68 | 68
  Apo-B | 8 (16) | -24 (18)

ADVERSE EVENTS:
Groups:
- Moxifloxacin: 400 mg Moxifloxacin: Positive control, unblinded treatment administered orally once during 1 of 3 crossover periods. There was at least 14 days washout between consecutive dosing periods.
Arm/Group | LY2484595 | Placebo | Moxifloxacin
Serious Adverse Events (participants affected / at risk) | 0/70 | 1/69 | 0/69
Other Adverse Events (participants affected / at risk) | 33/70 | 24/69 | 11/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2484595 (N=70) | Placebo (N=69) | Moxifloxacin (N=69)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2484595 (N=70) | Placebo (N=69) | Moxifloxacin (N=69)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (2) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 14 (16) | 4 (4) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Application site dermatitis (General disorders) | 2 (2) | 1 (1) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Application site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Application site rash (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (7) | 4 (4) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Bladder dilatation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days